CLINICAL TRIAL: NCT06052280
Title: Management of Initial Parkinson's Disease: a Prospective, Mono-centric, no Profit Pilot Clinical Trial Comparing Conventional Face-to-face Physiotherapy and Home-based Telerehabilitation
Brief Title: Pilot Study: Parkinson's Conventional Physiotherapy vs Home-based Telerehabilitation
Acronym: PD-REHAB-NET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale CN1 Cuneo (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resolution 982 of May 16, 2023
Record Dates: First submitted 2023-09-11; First posted 2023-09-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Telerehabilitation; Physical Activity; Physical Therapy Modalities
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This pilot study is designed to assess the feasibility of the integrated multidimensional approach in treating and rehabilitating PD patients in a local clinical setting, both for the Telerehabilitation Exercise (TrE) arm and for the Home Self-Exercise (HSE) arm, by:
  1. assessing participants' inclusion/exclusion criteria, testing instruments/procedures, testing data collection method;
  2. obtaining preliminary data to estimate sample size for the primary outcome, in both arms;
  3. evaluating appropriateness of the consent form, recruitment potentials, and the required number of researchers needed for study management;
  4. assessing patients' acceptability of the intervention and their compliance. Secondary objectives are the monitoring of patients' perceived quality of life, and of motor performance and non-motor symptoms through specific rating scales.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Exercise group (TrE arm) (Experimental)
  Interventions: Other: Telerehabilitation exercise program
- Home Self-Exercise group (HSE arm) (Active Comparator)
  Interventions: Other: Home self-exercise program

INTERVENTIONS:
Other: Telerehabilitation exercise program — After the outpatient intensive physical therapy program (common to both study arms), patients in the TrE group will continue with prescribed self-training at home through telerehabilitation, at least 3 times a week for 4 weeks. Each physical exercise session will consist of at least 5 minutes of aerobic warming-up, 35 minutes of specific high-intensity exercises for PD, and 5 minutes of aerobic cool-down.
  The TrE arm will be supported by a telerehabilitation device which will be installed and tested at the patients' home immediately after the outpatient intensive program. The device will track any access and exercise duration, so that the physiotherapists will be able to remotely monitor both the actual duration of each session and their weekly frequency. One session per week will be directly and online supervised by a physiotherapist, while the other two will be recorded only.
  Other Names: Virtual self-exercise program
  Arms: Telerehabilitation Exercise group (TrE arm)
Other: Home self-exercise program — After the outpatient intensive physical therapy program (common to both study arms), patients in the HSE group will continue with prescribed self-training at home, at least 3 times a week for 4 weeks. Each physical exercise session will consist of at least 5 minutes of aerobic warming-up, 35 minutes of specific high-intensity exercises for PD, and 5 minutes of aerobic cool-down.
  The HSE arm will be given a booklet containing detailed explanations and pictures of the assigned exercises, in order to guide them in the correct execution of the requested movements. Subjects in this group will be asked to fill in a training diary to keep track of the training sessions and their duration. Once a week a physiotherapist will contact patients to discuss possible problems encountered in performing the exercises and to help in solving them.
  Other Names: Conventional self-exercise program
  Arms: Home Self-Exercise group (HSE arm)

SUMMARY:
The Parkinson TELEREHABilitation-NET pilot study (Parkinson TELEREHAB-NET) is designed to observe and monitor PD patients in their initial phase (which includes the period from the onset of motor symptoms until the onset of motor fluctuations) and to assess the feasibility of an integrated multidimensional approach in treating and managing PD patients in a local clinical setting (ASL CN1). Chiefly, through this pilot study, feasibility and acceptability of the general experimental plan, as well as the potential for positive effects of physiotherapy in early PD patients will be assessed.

So, this pilot study primarily aims at:

1. validating the feasibility of the study protocol, assessing participants' inclusion and exclusion criteria, testing instruments/procedures used for home rehabilitation (both for the Telerehabilitation Exercise group - TrE arm and for the Home Self-Exercise group - HSE arm), testing the suitability of the method for data collection;
2. obtaining the required preliminary data for the calculation of a sample size for the primary outcome, in both arms;
3. evaluating appropriateness of the consent form, recruitment potentials, time needed to receive written consent, and the required number of researchers/medical specialists/physiotherapists needed to cover the whole study path;
4. assessing patients' acceptability of the intervention, through the evaluation of the adherence to rehabilitation process (in both arms), the completeness of proposed measurements, and compliance at follow-up.

Secondary objectives are the monitoring of patients' perceived quality of life, and of motor performance and non-motor symptoms through specific rating scales, after completing the whole rehabilitation path (described below) compared to baseline level, and maintenance of results over time.

ELIGIBILITY:
Inclusion Criteria:

General:

* adults, aged 18 or older;
* medical diagnosis of idiopathic PD according the most recent Movement Disorder Society diagnostic criteria;
* disease stage ≤ 2 on the Hoehn&Yahr scale;
* Montreal Cognitive Assessment score >25;
* ability to read, understand and provide a written informed consent, in accordance with good clinical practice and local regulations;
* motivation and possibility to show up for planned controls and to comply with the requested study procedures.

Specific for TrE arm:

* wireless internet access at home;
* adequate room to place telerehabilitation device (about 2 meters in front of device monitor).

Exclusion Criteria:

* <18 years of age;
* Any atypical, iatrogenic, or secondary Parkinsonism;
* Disease stage > 2 on the Hoehn&Yahr scale;
* Any severe orthopaedic, vascular, respiratory, or cardiac problems or any other medical condition that, in the principal investigator's opinion, could limit participation in moderate exercise or the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Study recruitment potentials | baseline
  total number of enrolled subjects / total number of eligible subjects
Single arm recruitment potentials | baseline
  arm-specific number of enrolled subjects / arm-specific number of eligible subjects
Adherence to study path | at end of outpatient intensive exercise program (4 weeks from baseline), after training at home (8 weeks from baseline), and for home-based training (follow-ups at 6 months and at 12 months from baseline)
  drop-out rate at each single step, total and by arm
Compliance to interventions | at end of outpatient intensive exercise program (4 weeks from baseline), after training at home (8 weeks from baseline), and for home-based training (follow-ups at 6 months and at 12 months from baseline)
  number of fulfilled visits / number of scheduled visits

SECONDARY OUTCOMES:
Cognitive functions | from baseline to follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Montreal Cognitive Assessment. This scale ranges from 0 to 30 points, with higher scores meaning a better outcome.
Freezing of gait | from baseline to follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Freezing of Gait Questionnaire. This scale ranges from 0 to 24 points, with higher scores meaning a worse outcome.
Movement disorders | from baseline to follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Movement Disorder Scale (parts 1, 2, 3, and 4). This scale ranges from 0 to 260 points, with higher scores meaning a worse outcome.
Postural control | from baseline to follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Mini-Balance Evaluation System Test. This scale ranges from 0 to 28 points, with higher scores meaning a better outcome.
Sensory orientation | from baseline to follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Non-Motor Symptom Scale. This scale ranges from 0 to 360 points, with higher scores meaning a worse outcome.
Quality of life perception | from baseline to follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Parkinson's Disease Quality of Life Questionnaire. This scale ranges from 0 to 32 points, with higher scores meaning a worse outcome.
Walking ability | after active interventions (at 4 weeks and at 8 weeks from baseline) and at follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in 6-minute walking test. This test measures how many meters the patient can cover in 6 minutes. The minimum is 0 meter, the maximum is not pre-specified; a longer distance means a better outcome.
Transition ability between sitting and standing | after active interventions (at 4 weeks and at 8 weeks from baseline) and at follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in 5-time sit-to-stand test. This test measures in how many seconds the patient manages to sit and stand for 5 times. Minimum and maximum time lengths are not pre-specified; a higher time means a worse outcome.
Backward walking ability | after active interventions (at 4 weeks and at 8 weeks from baseline) and at follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in 3-meter backward walking test. This test measures in how many seconds the patient manages to walk backward for a 3 meters distance. Minimum and maximum time lengths are not pre-specified; a higher time means a worse outcome.
Turning ability | after active interventions (at 4 weeks and at 8 weeks from baseline) and at follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in 360° turn right-to-left test. This test measures in how many seconds the patient manages to perform a complete 360° turn from right to left. Minimum and maximum time lengths are not pre-specified; a higher time means a worse outcome.
Manual dexterity | after active interventions (at 4 weeks and at 8 weeks from baseline) and at follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Coin rotation test. This test measures how many times the patient manages to turn a coin (of 25 millimeters in diameter) in 30 seconds. The minimum is 0, the maximum is not pre-specified; more the times better the outcome.
Transition ability between standing and prone position | after active interventions (at 4 weeks and at 8 weeks from baseline) and at follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in Stand-prone-stand test. This test measures in how many seconds the patient takes to change position from standing to prone to standing again. Minimum and maximum time lengths are not pre-specified; a higher time means a worse outcome.
Dynamic stability | after active interventions (at 4 weeks and at 8 weeks from baseline) and at follow-ups (at 6 months and at 12 months from baseline)
  Possible patients' changes in 4-square-step test. This test measures in how many seconds the patient sequentially steps over four delimited areas (1 square meter large). Minimum and maximum time lengths are not pre-specified; a higher time means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elona Brahimi, MD, Principal Investigator — Neurology Unit, Movement Disorders Clinic , Local Health Authority, ASL Cuneo 1, Italy
Locations (1):
- Azienda Sanitaria Locale CN1, Cuneo, Italy

IPD SHARING:
Plan to Share IPD: No